CLINICAL TRIAL: NCT05425485
Title: educAR: Validation of a Double Educational Strategy to Improve Therapeutic Adherence in Rheumatoid Arthritis.
Brief Title: educAR: Improving Adherence in Rheumatoid Arthritis
Acronym: educAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: María Ahijón (Other)
Collaborators: Instituto de Salud Musculoesquelética SL (Unknown)
Responsible Party: Sponsor-Investigator, María Ahijón, Principal investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4710
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Therapeutic adherence; Patient education
MeSH Terms: conditions — Arthritis, Rheumatoid; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Cluster-trial
Who Masked: Participant
Masking Description: The patients are invited to participate in an observational study of adherence, as the intervention is done at the level of the care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EducAR strategy (Active Comparator): Healthcare personnel involved in the care of patients with RA in the selected centres will be provided with access to a website and instructed in its use in a videoconference. The website includes a training section for healthcare professionals and another for patients. The former includes explanatory videos on how to manage doctor-patient communication and to facilitate adherence and what not to do, tools to explain treatment options (shared decision aids) and links to key documents. The patient section includes information for patients (downloadable in leaflet format), medication calendars and disease diaries, videos explaining medication administration in RA and links to patient associations, among other tools.
  Both access to the website and its materials and to the instruction session will be open to all those involved in the corresponding service, but will not be mandatory.
  Interventions: Behavioral: Multi-component intervention
- Standard of care (No Intervention): Physicians in the control group will not be instructed and will have no access to the materials included in the physician section of the webpage.

INTERVENTIONS:
Behavioral: Multi-component intervention — Web-based strategy with processes, materials, and patient and doctor education formats.
  Other Names: EducAR
  Arms: EducAR strategy

SUMMARY:
Based on recent guidelines, the investigators have developed a parallel (patient and physician) educational web-based tool. To prove its effectiveness, the investigators have designed a cluster clinical trial of a 6-month duration in which 15 centres will be randomised to receive access and instruction on the strategy or to continue standard care.

The trial endpoint is adherence at the patient level, for which each centre will recruit 15 consecutive patients and measure adherence (medication, physical activity, Mediterranean diet) and disease activity as of baseline and 6 months after.

DETAILED DESCRIPTION:
Treatment adherence in patients with rheumatoid arthritis (RA) is estimated to be between 50-80%. Non-adherence is a health problem with a significant economic impact. The causes of non-adherence are multiple and require individualized care that is difficult both to implement at the professional level and to prove effective.

Based on recent international recommendations and previous work from the research team, plus a qualitative study with multi-stakeholders, the investigators have designed a web-based strategy to avoid non-adherence in RA.

The primary objective is to evaluate the effectiveness of an evidence-based, consensus-based adherence intervention strategy for improving adherence in patients with RA.

Secondary objectives are to evaluate the impact on disease activity, healthy habits (diet/exercise), cardiovascular risk factors, quality of life and patient satisfaction.

The investigators have designed a cluster clinical trial of 6-month duration.

Fifteen centres will be randomised to receive access and instruction on the strategy or to continue standard care. Centre recruitment is on a voluntary basis, understanding that access to the educational tool will be delayed in case of being assigned to the control group.

The intervention is a web-based tool with educational and practical materials for the patient and for the physician (this part will be protected with a password during the duration of the trial). Physicians (prescribers or non-prescribers) in centres assigned to the intervention will be invited to be instructed on the materials (text, videos, checklists, calendars, etc).

Control will be standard care.

Each centre will recruit 15 consecutive adult patients with rheumatoid arthritis (as stated in the clinical records), less than 2 years since diagnosis and living independently.

The primary outcome will be therapeutic adherence (patient-level), defined as a score ≥ 80% in the Compliance Questionnaire on Rheumatology (CQR) and in the Adherence Medication Scale (RAM).

Secondary outcomes will be adherence to physical activity, a Mediterranean diet, lifestyle changes and disease activity.

Accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 79 patients per group are required, assuming that the initial proportion of adherent patients is 70% and at the end of the intervention, it would increase to 90% (only in the intervention group, in the control it would not change). A lost-to-follow-up rate of 25% has been estimated.

If 10 centres are selected to have at least 5 clusters for each group, this would correspond, rounding up, to 16 patients per centre, or a total of 160 patients.

The effect of the intervention on adherence to treatment will be refuted by the chi-square test and measured by relative risk (RR) and difference of proportions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* RA according to diagnosis recorded in clinical records
* < 2 years since diagnosis of rheumatoid arthritis.
* Independent daily living.

Exclusion Criteria:

* Cognitive impairment
* Language barriers
* Impossibility of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with therapeutic adherence. | 6 months
  Score ≥ 80% both in the Compliance Questionnaire in Rheumatology (CQR) plus the in Adherence Medication Scale (RAM).

SECONDARY OUTCOMES:
Adherence to physical exercise | 6 months
  Measured using the Exercise Attitude Questionnaire-18 (EAQ-18). Final result is expressed out of 100 point. High scores indicate great adherence to exercise.
Adherence to mediterranean diet | 6 months
  Measured using the Mediterranean Diet Adherence Screener (MEDAS).Patients with a score <9 will be considered poor adherents to the Mediterranean diet.
Disease activity | 6 months
  Measured using disease activity score of 28 joints (DAS28-ESR).This index stratifies disease activity into: high (>5.1), moderate (3.2-5.1), low (2.6- <3.2) and remission (<2.6).
Degree of satisfaction with medical care | 6 months
  Measured using the Arthritis Satisfaction questionnaire. Final result is expressed in a range from 0 to 100 points. Higher scores indicate greater satisfaction.
Health-related quality of life measured using the Short-form12 (SF-12) version 2 questionnaire, a shortened version of the SF-36 | 6 months
  Measured with the SF-12 version 2. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Overall Officials: María Ahijon, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (15):
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario de Elda, Elda
  - Hospital Universitari d'Igualada, Igualada
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital de la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Ahijon Lana M, Sivera Mascaro F, Fernandez-Nebro A, Muntadas Castello S, Perez M, Oton T, Garcia de Yebenes MJ, Carmona L; EDUCAR Group. EducAR: implementing a multicomponent strategy to improve therapeutic adherence in rheumatoid arthritis. RMD Open. 2025 Feb 27;11(1):e004989. doi: 10.1136/rmdopen-2024-004989. PMID 40021204

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT05425485/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT05425485/ICF_001.pdf